CLINICAL TRIAL: NCT06606743
Title: The Comparative Impacts of High-Intensity Interval Training and Power Training on Heart Rate Variability, Gait, and Functional Performance in Patients With Parkinson's Disease
Brief Title: Interval Training and Parkinson's Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Miami (Other)
Responsible Party: Principal Investigator, Joseph Signorile, Professor, University of Miami
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20240865
Record Dates: First submitted 2024-09-16; First posted 2024-09-23 (Actual); Last update posted 2025-08-15 (Actual); Status verified 2025-08

CONDITIONS: Other Disorders of Autonomic Nervous System
Keywords: Interval Training; Resistance Training
MeSH Terms: interventions — High-Intensity Interval Training

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High-Intensity Interval Training (Experimental): Participants in this group will receive high-intensity interval training 2 times per week for 10 consecutive weeks.
  Interventions: Behavioral: High-Intensity Interval Training
- High-Velocity Circuit Resistance Training (Active Comparator): Participants in this group will receive high-velocity circuit resistance training 2 times per week for 10 consecutive weeks.
  Interventions: Behavioral: High-Velocity Circuit Resistance Training

INTERVENTIONS:
Behavioral: High-Intensity Interval Training — Participants will receive a total of 20 in-person sessions of 45 minutes duration. Subjects perform high-speed movements with minimal recovery between movements. Hand weight will be used to increase intensity as training progresses.
  Arms: High-Intensity Interval Training
Behavioral: High-Velocity Circuit Resistance Training — Participants in this group will perform a total of 20 in-person training sessions using 12 resistance exercises performed in 3 circuits with minimal recovery between exercises.
  Arms: High-Velocity Circuit Resistance Training

SUMMARY:
This research is designed to compare the impact of high-intensity interval training and high-velocity circuit resistance training on heart rate variability, gait, and functional performance in patients with Parkinsons disease.

ELIGIBILITY:
Inclusion Criteria:

1. Confirmed diagnosis of Parkinson's disease
2. Between the ages of 30-90 years of age;
3. Movement Disorder Society-Unified Parkinson's Disease Rating Scale ≤2, which will be provided by the participant's medical provider and be evaluated within 1 year of the study's inception.

Exclusion Criteria:

1. Uncontrolled cardiovascular disease that prevents participation in a training program
2. Documented HIV infection or another immunodeficiency syndrome
3. Other neuromuscular diseases besides Parkinson's disease
4. Current musculoskeletal injury that prevents exercise.
5. Having a pacemaker or other internal medical devices

Ages: 30 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2024-09-20 (Actual); Primary Completion 2025-06-30 (Actual); Study Completion 2025-06-30 (Actual)

PRIMARY OUTCOMES:
Changes in Heart Rate Variability | Baseline, 10 weeks
  After a 10-minute supine rest on a padded treatment table, subjects will breathe at a rate of six breaths per minute for two minutes. The heart rate will be monitored using a Polar heart rate monitor and variations will be detected using the elite application via mobile device.
Changes in the Six-Minute Walk Test | Baseline, 10 weeks
  The objective of the test is to walk as far as possible for six minutes. The subject will walk at a normal pace around a marked course for six minutes. The subject may stop to rest and begin again at will. The distance covered indicates aerobic fitness. The further a person walks, the better their cardiovascular condition. The units are meters.
Changes in the Ten-Meter Walk Test | Baseline, 10 weeks
  The ten-meter walk test will be used to assess gait velocity. The participants will be asked to walk as quickly as possible in a straight line on a 10-m course marked at 0, 2, 8 and 10 m. On verbal command, participants will start on the 0-m mark and stop when they cross the 10-m mark. The total time to ambulate from the 2-m mark to the 8-m mark (6 m total) will be timed to the hundredth of a second. Two trials will be performed, and the average will be documented in meters per second. One-minute recoveries will be provided between trials. Total time is 420 seconds.
Changes in the Five Times Sit-to-Stand Test | Baseline, 10 weeks
  The five time sit-to-stand test will be used to assess functional lower body strength. The participant will sit with their arms folded across their chest and their back against the chair. On verbal command, the participant will stand up and sit down 5 times as quickly as possible. Timing begins at "Go" and ends when the buttocks touch the chair after the 5th repetition. One practice and two testing trials will be performed. Time will be measured in seconds.
Changes in Heart Rate Recovery | Baseline, 10 weeks
  Following the Six-Minute Walk Test, participants will be asked to sit quietly for one-minute and heart rate recovery will be determined by analyzing the participant's heart rate immediately following the Six-Minute Walk Test and again after the one-minute recovery. The difference in beats between the two times will be calculated and used for analysis
Changes in One Repetition Maximum Strength | Baseline, 10 weeks
  A one-repetition maximum test measures the maximum load that an individual can lift only a single time throughout the full range of motion of the chest press and leg press exercises using proper form. All subjects' one-repetition maximum values will be determined within four to five trials. The units of measure are kilograms. Testing is performed on computerized, pneumatic machines.
Changes in Neuromuscular Power Testing | Baseline, 10 weeks
  Peak muscle power is then measured at eight relative intensities (40, 50, 60, 70, and 80% of one repetition maximum) on the computerized pneumatic machines. For each repetition, the concentric phase is performed as fast as possible, and the eccentric phase lasts between 2 and 3 seconds. Power testing is done for the leg press and chest press, and the unit of measurement is Watts.
Changes in Swing time of Gait | Baseline, 10 weeks
  Movement analyses will be performed during the ten-meter walk test. The measure will be swing time. Swing time is how long it takes to swing the back foot forward to initiate a new step. The unit of measurement is seconds.
Changes in Stance Time of Gait | Baseline, 10 weeks
  Movement analyses will be performed during the ten-meter walk test. The measure will be stance time. Stance time is the duration of the time between heel strike and toe off of the same foot. The unit of measurement is seconds.
Changes in Double Support time of Gait | Baseline, 10 weeks
  Movement analyses will be performed during the ten-meter walk test. The measure will be double support time. Double support time is how long both feet are in contact with the ground. The unit of measurement is seconds.
Changes in Step Time of Gait | Baseline, 10 weeks
  Movement analyses will be performed during the ten-meter walk test. The measure will be step time. Step time is how long one foot is in contact with the ground. The unit of measurement is seconds.
Changes in Cadence of Gait | Baseline, 10 weeks
  Movement analyses will be performed during the ten-meter walk test. The measure will be cadence. Cadence is the number of steps per minute. The unit of measurement is steps per minute.
Changes in Stride Length of Gait | Baseline, 10 weeks
  Movement analyses will be performed during the ten-meter walk test. The measure will be stride length. Stride length is the distance covered when a person takes two steps. The unit of measurement is meters.
Changes in Step Length of Gait | Baseline, 10 weeks
  Movement analyses will be performed during the ten-meter walk test. The measure will be step length. Step length is the distance covered when a person takes one step. The unit of measurement is meters.
Changes in speed of Gait | Baseline, 10 weeks
  Movement analyses will be performed during the ten-meter walk test. The measure will be speed. Gait speed is how fast a person walks. The unit of measurement is meters per second.
Changes in Stride Width of Gait | Baseline, 10 weeks
  Movement analyses will be performed during the ten-meter walk test. The measure will be stride width. Stride width is the side-to-side distance between the line of the two feet during gait. The measurement is in meters.

SECONDARY OUTCOMES:
Changes in the Parkinson's Disease Questionnaire-39 | Baseline, 10 weeks
  The Parkinson's Disease Questionnaire-39 is a 39-item self-report questionnaire that assesses Parkinson's disease-specific health-related quality over the last month across the eight quality of life dimensions and specific dimensions of functioning and well-being. Each question is scored from 0-4 points, with lower scores reflecting better quality of life.
Non-Motor Symptoms Scale for Parkinson's Disease | Baseline, 10 weeks
  The Non-Motor Symptoms Scale for Parkinson's Disease is a 30-item validated and reliable measure of non-motor symptoms that many patients with Parkinson's Disease experience. The scale is grouped into nine domains including cardiovascular, sleep/fatigue, attention/memory, gastrointestinal, urinary, sexual function, perceptual problems/hallucinations, mood/cognition, and miscellaneous. The score is based on the degree of severity (from 0-3) and frequency (from 1-4). The test is administered by a healthcare professional in an interview format.

CONTACTS AND LOCATIONS:
Overall Officials: Joseph F. Signorile, PhD, Principal Investigator — University of Miami
Locations (2):
- United States (2):
  - University of Miami, Coral Gables, Florida
  - Laboratory of Neruomuscular Research and Active Aging, Coral Gables, Florida

IPD SHARING:
Plan to Share IPD: No